CLINICAL TRIAL: NCT01013545
Title: Developmental and Augmented Intervention for Facilitating Expressive Language
Acronym: CCNIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Autism Speaks (Other)
Collaborators: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); Vanderbilt University (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Principal Investigator, Professor, Ph.D., Autism Speaks
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G09-04-013-01; 5666 (Other Grant/Funding Number: Autism Speaks)
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Joint Engagement + Enhanced Milieu Training; Joint Engagement + Enhanced Milieu Training+Augmentative Communication (AAC)
Keywords: joint engagement; augmentative communication (AAC); enhanced milieu training; autism spectrum disorder; language
MeSH Terms: conditions — Autism Spectrum Disorder; Language

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JAE-EMT (Experimental): The interventionist will coach the caregiver and child while they engage in play routines established through collaboration between caregiver and interventionist. This intervention condition uses spoken language as the mode of communication. Individual, single word targets will be selected based on the child's level of language production and specific interests. The targets are systematically modeled in response to child actions and attention during play. A sequence of milieu teaching prompts will also be used to elicit targets from the child when use of the target language is functional for the child.
  Interventions: Behavioral: JAE Intervention
- JAE-AAC (Experimental): The interventionist will coach the caregiver and child while they engage in play routines established through collaboration between caregiver and interventionist. The mode of communication introduced in this intervention condition is a developmentally chosen augmentative communication device. These devices are provided with a set of individually selected visual-graphic symbols and a relevant lexicon. The use of the device is taught within natural communicative exchanges within play routines and daily activities.
  Interventions: Behavioral: JAE Intervention

INTERVENTIONS:
Behavioral: JAE Intervention — The overall goal in each session will be for the caregiver-child dyad to be in a state of supported or coordinated joint engagement. In this state the child is aware of the other's activity, and may actively coordinate their attention between an object/toy and the caregiver. The interventionist will coach the caregiver and child while they engage in play routines established through collaboration between caregiver and interventionist.

SUMMARY:
This study will contrast two experimental treatment conditions by testing whether joint attention/joint engagement intervention using spoken communication (JAE-EMT) results in better outcomes than joint attention/joint engagement intervention that is instead supplemented with an individualized AAC system (JAE-AAC). Thus, the skills of joint attention/joint engagement (JAE) remain foundational to developing expressive language but the difference in the two treatments will be between whether the JAE is administered through the more traditional spoken means (EMT) or through an augmentative and alternative communication device (AAC).

DETAILED DESCRIPTION:
Both treatments will be manualized and a novel research design method called Sequential Multiple Assignment Randomized Trial (SMART) will be applied. SMART design will allow the interventionists to adjust the course of treatment based on whether the children respond to the treatment. More specifically, there will be two stages of intervention and during Stage 1, 90 nonverbal (e.g. those who have less than 5 spoken words) children with ASD between 5 and 8 years of age will be randomly assigned to either the JAE-EMT or JAE-AAC group. After receiving the assigned Stage 1 treatment for 12 weeks, all participants will be assessed to see if they responded to the Stage 1 treatment. If the children do respond to Stage 1 treatment, they will continue with that same treatment for another 12 weeks in Stage 2. A different treatment sequence will be used for those who do not respond to Stage 1 treatment where these non-responders will be re-assigned to 1 of 3 alternative intervention conditions. For example, those who do not respond to JAE-AAC will have the intensity of that same JAE-AAC treatment increased. Those who do not respond to the other, JAE-EMT treatment will be randomly assigned to either a more intense JAE-EMT condition, or the original JAE-AAC implemented in Stage 1. At the end of Stage 2, another follow-up assessment of cognitive, language, and social communication skills will be administered. Furthermore, several children who enter the study in the early stages will be tested again, 3 months after the Stage 2 follow up (not all children will be able to be tested at 9 months within the 3 year grant period).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism from a licensed psychologist or board certified developmental pediatrician, or child and adolescent psychiatrist, confirmed by Module 1 of the Autism Diagnostic Observation Schedule (Lord et al., 2001)
* Chronological age between 5 and 8 years
* Classified as nonverbal with fewer than 20 spontaneous expressive words as determined by parent report, language sample, and standardized tests.
* Demonstrated slow or no progress in expressive language acquisition despite at least 2 years of early intervention

Exclusion Criteria:

* Major medical conditions other than autism, specifically: a) motor disabilities such as cerebral palsy or tuberous sclerosis, b) sensory disabilities such as blindness or deafness, and c) genetic disorders such as Fragile X or Down syndrome.
* Nonverbal mental age < 24 months, based on a nonverbal score from the Leiter-R (Roid & Miller, 1997).

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of words used spontaneously during language sample | 3 months
  Change in spontaneous language from beginning of treatment, to the mid-point.

SECONDARY OUTCOMES:
Number of words used spontaneously during language sample | 6 months
  Change in spontaneous language used at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Connie Kasari, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Background] Kasari C. Assessing change in early intervention programs for children with autism. J Autism Dev Disord. 2002 Oct;32(5):447-61. doi: 10.1023/a:1020546006971. PMID 12463519
- [Background] Kasari C, Paparella T, Freeman S, Jahromi LB. Language outcome in autism: randomized comparison of joint attention and play interventions. J Consult Clin Psychol. 2008 Feb;76(1):125-37. doi: 10.1037/0022-006X.76.1.125. PMID 18229990
- [Background] Kasari C, Freeman S, Paparella T. Joint attention and symbolic play in young children with autism: a randomized controlled intervention study. J Child Psychol Psychiatry. 2006 Jun;47(6):611-20. doi: 10.1111/j.1469-7610.2005.01567.x. PMID 16712638
- [Background] Millar DC, Light JC, Schlosser RW. The impact of augmentative and alternative communication intervention on the speech production of individuals with developmental disabilities: a research review. J Speech Lang Hear Res. 2006 Apr;49(2):248-64. doi: 10.1044/1092-4388(2006/021). PMID 16671842
- [Background] Kaiser AP, Trent JA. Communication intervention for young children with disabilities: Naturalistic approaches to promoting development. In S Odom, R Horner, M Snell & J Blacher (Eds), Handbook of Developmental Disabilities. New York: Guilford Press, 2007.
- [Background] Kaiser AP, Hancock TB, Nietfeld, JP. The effects of parent-implemented enhanced milieu teaching on the social communication of children who have autism. Journal of Early Educaiton and Development [Special Issue] 4: 423-446, 2000.
- [Background] Landa R. Early communication development and intervention for children with autism. Ment Retard Dev Disabil Res Rev. 2007;13(1):16-25. doi: 10.1002/mrdd.20134. PMID 17326115
- [Background] Hancock TB, Kaiser, AP. Enhanced Milieu Teaching. In R. McCauley & M. Fey (Eds.) Treatment of language disorders in children. Baltimore: Paul H. Brookes. 2006.
- [Result] Shire SY, Goods K, Shih W, Distefano C, Kaiser A, Wright C, Mathy P, Landa R, Kasari C. Parents' Adoption of Social Communication Intervention Strategies: Families Including Children with Autism Spectrum Disorder Who are Minimally Verbal. J Autism Dev Disord. 2015 Jun;45(6):1712-24. doi: 10.1007/s10803-014-2329-x. PMID 25475363
- [Result] Kasari C, Patterson S. Interventions addressing social impairment in autism. Curr Psychiatry Rep. 2012 Dec;14(6):713-25. doi: 10.1007/s11920-012-0317-4. PMID 23055002
- [Derived] Almirall D, DiStefano C, Chang YC, Shire S, Kaiser A, Lu X, Nahum-Shani I, Landa R, Mathy P, Kasari C. Longitudinal Effects of Adaptive Interventions With a Speech-Generating Device in Minimally Verbal Children With ASD. J Clin Child Adolesc Psychol. 2016 Jul-Aug;45(4):442-56. doi: 10.1080/15374416.2016.1138407. Epub 2016 Mar 8. PMID 26954267
- [Derived] Kasari C, Kaiser A, Goods K, Nietfeld J, Mathy P, Landa R, Murphy S, Almirall D. Communication interventions for minimally verbal children with autism: a sequential multiple assignment randomized trial. J Am Acad Child Adolesc Psychiatry. 2014 Jun;53(6):635-46. doi: 10.1016/j.jaac.2014.01.019. Epub 2014 Mar 12. PMID 24839882